CLINICAL TRIAL: NCT03789851
Title: Minimally Invasive Biopsy Technique Predicting Breast Pathological Complete Respons After Neoadjuvant Chemotherapy for Breast Cancer
Brief Title: Minimally Invasive Biopsy Predicting Breast pCR After NAC for Breast Cancer
Acronym: MIBPBPCR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Director of the Breast Cancer Center, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MIB001
Record Dates: First submitted 2018-12-27; First posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy, Large-Core Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- core needle biopsy (Experimental): All patients enrolled in this study received a ultrasound-guided multipoint core needle biopsy after surgery.
  Interventions: Device: core needle biopsy

INTERVENTIONS:
Device: core needle biopsy — Because the ultrasound was unable to accurately position the marker clip, I125 coud be placed at the position of the marker clip under the guidance of preoperative mammography. The gamma detector was used to locate the tumor bed to guide the ultrasound-guided multi-point CNB. Ultrasound-guided multipoint CNB was used directly after breast conserving surgery or mastectomy. Centering on the marker clip, the range of 0.5 cm was the first area, and then the range of 0.5 cm was the second area, and so on, until the extent of the expansion reached the long diameter of the original tumor, and 4 pieces were uniformly taken in each area.
  Other Names: ultrasound-guided multipoint core needle biopsy

SUMMARY:
Neoadjuvant chemotherapy (NAC) is widely used as an efficient breast cancer treatment. Ideally, a pathological complete remission (pCR) can be achieved. With improvements in molecular typing guided NAC and targeted therapies, there has been dramatic improvement in pCR rates, especially among triple-negative and human epidermal growth factor receptor 2 positive breast cancers. Rates of pCR in these groups of patients can reach 60% or higher. NAC has significantly promoted the loco-regional de-escalating treatment of breast cancer, and the need for breast surgery in NAC cases with pCR has been questioned, especially in patients undergoing breast-conserving surgery with whole breast radiotherapy. The main impediments for potential elimination of breast surgery have been the fact that conventional and functional breast imaging techniques are incapable of accurate prediction of residual disease. However, imaging-guided minimally invasive biopsy (MIB) techniques might have the potential to overcome this impediment.

The investigators design and begin a prospective one-armed clinical study to explore the accuracy of MIB in predicting breast pCR after NAC.

DETAILED DESCRIPTION:
In clinical routine surgical treatment follows the neoadjuvant chemotherapy (NAC). However, recent studies have demonstrated that shrinking tumors need less surgical treatment indicating that patients with pCR could potentially be spared of surgery in the future. However, up to now, prediction of pCR after NACT is only moderately accurate. This prospective, monocenter diagnostic trial aims to explore if minimal invasive biopsies (MIB) might overcome this diagnostic challenge.

From June 1st, 2017 to June 15th, 2019 the investigators performed ultrasound-guided multipoint core needle biopsy (CNB) on 50 breast cancer patients after NAC and directly after surgery. To analyse CNB pathologically results were categorized as follows: residual vital tumor cells (invasive, in situ, both, lymphangiosis carcinomatosous) present, (significant parts of) the tumor bed present, neither vital tumor cells nor (significant parts of) the tumor bed (indicating a non representative VAB). The results were compared to those of the pathological examination of surgical specimen.

ELIGIBILITY:
Inclusion Criteria:

* after full-course neoadjuvant chemotherapy (NAC) according to the NACT protocol
* with cT1c-cT4a-c tumors
* after informed consent
* with breast ultrasound, mammography (and breast MRI where necessary) before and after NACT
* Clinical / imaging partial or complete response to NAC
* Any routine breast cancer surgical intervention planned according to guidelines (breast conservation or mastectomy)
* Residual intramammary target lesion or clip marker is visible in ultrasound and / or mammography
* Inclusion of only one breast per patient, in bilateral cancer one breast can be included
* In case of multicentric disease: confirmation of the same tumorbiological subtype defined by immunohistology in at least 2 lesions.

Exclusion Criteria:

* Palliative or recurrent breast cancer
* Pregnancy and lactation
* cT4d stage (inflammatory breast cancer)
* M1 stages
* stable disease according to a multimodal assessment of ultrasound, mammography and breast MRI (if available) according to RECIST
* dislocation of marker (> 10mm distance to the initial lesion)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
false negative CNB results，reported as the false negative rate (= FNR) | after breast surgery, up to 2 weeks after CNB
  non-detected residual tumor by CNB (=index test) compared to breast surgery (=reference test): FNR = rate of patients with non-detected residual tumor by CNB compared to breast surgery Residual tumor is defined as a positive result; in surgical specimen as well as in CNB.

SECONDARY OUTCOMES:
negative predictive value (NPV) | after breast surgery, up to 2 weeks after CNB
  The negative predictive value (NPV) will be calculated as the quotient of the number of cases with pCR in CNB and in surgical specimen (= true negative result), divided by the total number of cases with pCR in CNB. Residual tumor is defined as a positive result; in surgical specimen as well as in CNB.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Cancer Center, Shandong Cancer Hospital Affiliated to Shandong University, Jinan, China